CLINICAL TRIAL: NCT05538195
Title: Chimeric Antigen Receptor T Lymphocytes (CAR-T) Targeting CEA in the Treatment of CEA Positive Clinical Study of Advanced Malignant Solid Tumors
Brief Title: Safety and Efficacy of CEA-targeted CAR-T for CEA-positive Advanced Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBC040
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-05

CONDITIONS: Gastric Cancer; Colon Cancer; Rectal Cancer; Esophageal Cancer; Pancreatic Cancer
MeSH Terms: conditions — Stomach Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous of CEA-targeted CAR-T (Experimental): Infusion of CEA-targeted CAR-T cells by dose of 3-10x10^6 cells/kg
  Interventions: Biological: CEA-targeted CAR-T cells
- intraperitoneal injection of CEA-targeted CAR-T (Experimental): Infusion of CEA-targeted CAR-T cells by dose of 1-10x10^6 cells/kg
  Interventions: Biological: CEA-targeted CAR-T cells

INTERVENTIONS:
Biological: CEA-targeted CAR-T cells — Administration method: intravenous infusion； Subjects will receive conditioning therapy by Fludarabine and Cyclophosphamide before cell infusion.
  Arms: Intravenous of CEA-targeted CAR-T
Biological: CEA-targeted CAR-T cells — Administration method: intraperitoneal injection；Subjects will receive conditioning therapy by Fludarabine and Cyclophosphamide before cell infusion.
  Arms: intraperitoneal injection of CEA-targeted CAR-T

SUMMARY:
This study is a single-arm, open-label, dose-escalating + dose-expansion clinical study, aiming to evaluate the safety and efficacy of CEA-targeted CAR-T cell preparations, and to preliminarily observe the study drug in CEA-positive advanced malignant tumors. The pharmacokinetic characteristics of CAR-T cell preparations for the treatment of patients with CEA-positive advanced malignancies were obtained and the recommended dose and infusion schedule.

DETAILED DESCRIPTION:
According to the different infusion methods, it is divided into two subgroups: intravenous infusion and local infusion through the peritoneal cavity. Each subgroup includes a dose exploration stage (Part A) and a dose expansion stage (Part B). 3 patients were explored, starting from the low-dose group, and in the dose expansion phase, the safety and efficacy were further verified according to the safe recommended dose obtained in the dose exploration phase.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female;
2. Advanced, metastatic or recurrent malignant tumors diagnosed by histology or pathology, mainly colorectal cancer, esophageal cancer, gastric cancer, and pancreatic cancer;
3. After receiving at least second-line standard treatment failure (disease progression or intolerance, such as surgery, chemotherapy, radiotherapy, etc.) or lack of effective treatment methods;
4. Immunohistochemical staining of tumor samples within 3 months confirmed that the tumor was CEA positive (clear membrane staining, positive rate ≥ 10%); , the positive rate ≥ 10%), the serum CEA of the patient is required to exceed 10ug/L.
5. At least one assessable lesion according to RECIST 1.1 criteria;
6. ECOG score 0-2 points;
7. No serious mental disorder;
8. Unless otherwise specified, the function of the vital organs of the subject shall meet the following conditions:

   1. Blood routine: white blood cells>3.0×10^9/L, neutrophils>0.8×10^9/L, lymphocytes cells>0.5×10^9/L, platelets>75×10^9/L, hemoglobin>80g/L;
   2. Cardiac function: echocardiography showed cardiac ejection fraction ≥50%, and no obvious abnormality was found on electrocardiogram;
   3. Renal function: serum creatinine≤2.0×ULN;
   4. Liver function: ALT and AST ≤3.0×ULN (for patients with liver tumor infiltration, it can be relaxed to ≤5.0×ULN);
   5. Total bilirubin≤3.0×ULN;
   6. Oxygen saturation ≥95% in non-oxygen state.
9. Have apheresis or venous blood collection standards, and have no other contraindications for cell collection;
10. Subjects agree to use reliable and effective contraceptive methods for contraception within 1 year after signing the informed consent form to receiving CAR-T cell infusion (excluding rhythm contraception);
11. The patients themselves or their guardians agree to participate in this clinical trial and sign the ICF, indicating that they understand the purpose and procedures of this clinical trial and are willing to participate in the research.

Exclusion Criteria:

1. Those who have central nervous system metastasis or meningeal metastasis at the time of screening are judged by the investigator to be unsuitable for inclusion;
2. Participated in other clinical studies within 1 month before screening;
3. vaccinated with live attenuated vaccine within 4 weeks before screening;
4. Received the following anti-tumor treatments before screening: Received chemotherapy, targeted therapy or other experimental drug treatments within 14 days or at least 5 half-lives (whichever is shorter);
5. Active infection or uncontrollable infection requiring systemic treatment;
6. Patients with intestinal obstruction, active gastrointestinal bleeding, or a history of gastrointestinal bleeding within 3 months;
7. Except for alopecia or peripheral neuropathy, the toxicity of previous anti-tumor therapy has not improved to the baseline level or ≤ grade 1;
8. Suffering from any of the following heart diseases:

   1. New York Heart Association (NYHA) stage III or IV congestive heart failure;
   2. Myocardial infarction or coronary artery bypass grafting (CABG) within 6 months before enrollment;
   3. Clinically significant ventricular arrhythmia, or a history of unexplained syncope (except those caused by vasovagal or dehydration);
   4. History of severe non-ischemic cardiomyopathy;
9. Patients with active autoimmune disease, or other patients requiring long-term immunosuppressive therapy;
10. Suffering from other uncured malignant tumors in the past 3 years or at the same time, except cervical carcinoma in situ and basal cell carcinoma of the skin;
11. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer test is greater than the normal range; hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C Virus (HCV) RNA test is greater than the normal range; human immunodeficiency virus (HIV) antibody positive; syphilis test positive;
12. Women who are pregnant or breastfeeding;
13. Other investigators deem it unsuitable to participate in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of CAR-T cell preparations in the treatment of CEA-positive advanced malignancies [Safety and Tolerability] | 1 month
  The incidence of adverse events after CEA CAR-T cell infusion was assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 5.0)
Obtained the recommended dose and infusion regimen of CAR-T cells for the treatment of patients with CEA-positive advanced malignancies[Safety and Tolerability] | 28 days
  Dose-limiting toxicity after CEA CAR-T cell infusion

SECONDARY OUTCOMES:
Assessing disease control rates of CAR-T cell preparations in CEA-positive advanced malignancies[Effectiveness] | 3 month
  Disease control rate: The proportion of subjects who achieved CR, PR, SD after CAR-T infusion accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
AUCS of CEA CAR-T cells [Cell dynamics] | 3 months
  AUCS is defined as the area under the curve in 90 days
CMAX of CEA CAR-T cells [Cell dynamics] | 3 months
  CMAX is defined as the highest concentration of CEA CAR-T cells expanded in peripheral blood
TMAX of CEA CAR-T cells[Cell dynamics] | 3 months
  TMAX is defined as the time to reach the highest concentration
Pharmacodynamics of CEA CAR-T cells[Cell dynamics] | 3 months
  The content of CEA in peripheral blood was detected by ELISA at the visit points specified in the research protocol

OTHER OUTCOMES:
Objective response rate (ORR) of CEA CAR-T treatment in patients with CEA-positive advanced malignancies[Effectiveness] | 1 years
  Objective response rate includes：The proportion of subjects who achieved CR, PR after CAR-T infusion accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
Duration of Response (DOR) of CEA CAR-T treatment in patients with CEA-positive advanced malignancies[Effectiveness] | 1 years
  DOR will be assessed from the first assessment of CR/PR/SD to the first assessment of recurrence or progression of the disease or death from any cause
Progress-free survival(PFS) of CEA CAR-T treatment in patients with CEA-positive advanced malignancies[Effectiveness] | 1 years
  PFS will be assessed from the first CEA-CAR-T cell infusion to death from any cause or the first assessment of progression(Assessed based on RECIST criteria)
Overall survival(OS)of CEA CAR-T treatment in patients with CEA-positive advanced malignancies[Effectiveness] | 1 years
  OS will be assessed from the first CEA-CAR-T cell infusion to death from any cause (Assessed by investigators based on IRECIST criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, MD, Principal Investigator — Henan Cancer Hospital
Locations (1):
- He'nan Cancer Hospital, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided